CLINICAL TRIAL: NCT07142434
Title: Neonatal Umbilical Catheter Pathway Simulator
Acronym: NeoPath
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, D ANDREA VITO, Medical Doctor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 7348
Record Dates: First submitted 2025-07-27; First posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Simulator Training; Neonates and Preterm Infants; Catherization

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- no-experienced neonatal ultrasound practitioners (Experimental): pratictioners who will test and validate the simulator.
  Interventions: Device: neonatal Umbilical Catheter Pathway Simulator

INTERVENTIONS:
Device: neonatal Umbilical Catheter Pathway Simulator — evaluate the quality of simulator

SUMMARY:
Currently, training for umbilical catheter placement in neonates is primarily focused on inserting the catheter into the umbilical vein. However, no models to date allow real-time ultrasound assessment of catheter tip navigation and final positioning during the procedure. This study introduces the first training simulator designed specifically to address this need, enabling operators to practice not only the insertion but also the ultrasonographic localization of the catheter tip during the placement process.

ELIGIBILITY:
Inclusion Criteria:

* Experts must have at least 3 years of experience in neonatal abdominal ultrasound or central line placement.

Trainees must be medical residents in their 3rd year or beyond.

Exclusion Criteria:

* Less than 3 years of relevant experience for expert participants. Less than 3rd year of specialty training for trainee participants.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2025-08-05 (Actual); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Neo Path | 12 months
  Evaluation of the simulator's practicality through a user satisfaction questionnaire.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Meinen RD, Bauer AS, Devous K, Cowan E. Point-of-care ultrasound use in umbilical line placement: a review. J Perinatol. 2020 Apr;40(4):560-566. doi: 10.1038/s41372-019-0558-8. Epub 2019 Nov 22. PMID 31758061
- [Result] Kaae R, Kyng KJ, Frederiksen CA, Sloth E, Rosthoj S, Kerrn-Jespersen S, Eika B, Sorensen JL, Henriksen TB. Learning Curves for Training in Ultrasonography-Based Examination of Umbilical Catheter Placement: A Piglet Study. Neonatology. 2020;117(2):144-150. doi: 10.1159/000503176. Epub 2019 Oct 29. PMID 31661695
- [Result] D'Andrea V, Prontera G, Rubortone SA, Pezza L, Pinna G, Barone G, Pittiruti M, Vento G. Umbilical Venous Catheter Update: A Narrative Review Including Ultrasound and Training. Front Pediatr. 2022 Jan 31;9:774705. doi: 10.3389/fped.2021.774705. eCollection 2021. PMID 35174113

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-11-20): https://cdn.clinicaltrials.gov/large-docs/34/NCT07142434/Prot_SAP_000.pdf